CLINICAL TRIAL: NCT06160466
Title: Assessing the Additional Neoplasia Yield of Computer-aided Colonoscopy in Follow-up Patients in a Screening Setting
Acronym: GENIAL-CO FU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NP4451
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-02

CONDITIONS: Colonic Adenoma; Adenoma; Polyp of Colon
Keywords: ADR; CADe; Follow-up
MeSH Terms: conditions — Adenoma; Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artificial intelligence arm Patients undergoing colonoscopy with artificial intelligence. (Experimental): Patients undergoing colonoscopy with artificial intelligence.
  Interventions: Device: CADe colonoscopy using GI Genius device
- Conventional Colonoscopy (Active Comparator): Standard Colonoscopy with white light
  Interventions: Device: White light

INTERVENTIONS:
Device: CADe colonoscopy using GI Genius device — We wanted to compare the diagnostic yield obtained by using CADe colonoscopy to the yield obtained by the standard colonoscopy (SC) in a follow-up pateints in the screening population.
  Arms: Artificial intelligence arm Patients undergoing colonoscopy with artificial intelligence.
Device: White light — White light endoscopy
  Arms: Conventional Colonoscopy

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic yield of CADe in a consecutive population undergoing colonoscopy. The main question it aims to answer is the Adenoma Detection Rate (ADR). Participants undergoing colonoscopy for follow-up in a screening setting will be randomized in a 1:1 ratio to either receive Computer-Aided Detection (CADe) colonoscopy or a conventional colonoscopy (CC). GI Genius is the AI software that will be used in the present trial and is intended to be used as an adjunct to colonic endoscopy procedures to help endoscopists to detect in real time mucosal lesions (such as polyps and adenomas, including those with flat (non-polypoid) morphology) during standard screening and surveillance endoscopic mucosal evaluations. It is not intended to replace histopathological sampling as a means of diagnosis.Researchers will compare the CADe group and the CC-group to see if CAD-e can increase the ADR significantly.

DETAILED DESCRIPTION:
en if colonoscopy is considered the reference standard for the detection of colonic neoplasia, polyps are still missed. In large administrative cohort or case-control studies, the risk of early post-colonoscopy cancer appeared to be independently predicted by a relatively low polyp/adenoma detection rate. The adenoma detection rate among different endoscopists has been shown to be strictly related with the risk of post-colonoscopy interval cancer. When considering the very high prevalence of advanced neoplasia in the FIT-positive enriched population, the risk of post-colonoscopy interval cancer due to a suboptimal quality of colonoscopy may be substantial. Available evidence justifies therefore the implementation of efforts aimed at improving adenoma detection rate, based on retraining interventions and on the adoption of innovative technologies, designed to enhance the accuracy of the endoscopic examination.Nowadays, Artificial intelligence (AI) is gaining increased attention and investigation, since it seems to improve the quality of medical diagnosis and treatment. In the field of gastrointestinal endoscopy, two potential roles of AI in colonoscopy have been examined so far: automated polyp detection (CADe) and automated polyp histology characterization (CADx). CADe can minimize the probability of missing a polyp during colonoscopy, thereby improving the adenoma detection rate (ADR) and potentially decreasing the incidence of interval cancer. GI Genius is the AI software that will be used in the present trial. The software is developed by Medtronic Inc. (Dublin, Ireland) and is intended to be used as an adjunct to colonic endoscopy procedures to help endoscopists to detect in real time mucosal lesions (such as polyps and adenomas, including those with flat (non-polypoid) morphology) during standard screening and surveillance endoscopic mucosal evaluations. It is not intended to replace histopathological sampling as a means of diagnosis.

The objective of this study was to compare the diagnostic yield obtained by using CADe colonoscopy to the yield obtained by the standard colonoscopy (SC). As the risk of progression is higher for large than for small adenomas the specific contribution of the new technique in reducing the miss rate of large neoplasms represents an important outcome to be assessed in the study. In addition, given the suggested association of a higher miss-rate of serrated and flat lesions with an increased risk of early post-colonoscopy CRC, the benefit of the new technique in reducing the miss rate of these lesions will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50 to 74 undergoing colonoscopy examination following a prior colonsocopy were polyps were found (follow-up) performed in the context of a regional mass-screening program.

Exclusion Criteria:

* Patients unwilling or unable to give informed consent.
* Patients reporting use of anti-platelet agents or anticoagulants precluding removal of polyps.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Rate of advanced adenomas | When available the histological report of polyps removed (up to 3 weeks).
  The percentage of patients with adenomas with high-grade displasia in CADe colonoscopy group will be recorded and compared with the rate of patients with adenomas with high-grade displasia in standard colonoscopy group.
Rate of patients detected with 3 or more adenomas. | When available the histological report of polyps removed (up to 3 weeks).
  The percentage of patients with 3 or more adenomas (serrated adenomas will also be considered in the calculation) in CADe colonoscopy group will be compared with the rate of patients with 3 or more adenomas (including serrated adenomas) in standard colonoscopy group.

SECONDARY OUTCOMES:
Overall adenoma and polyp detection rate, flat adenoma and serrated polyps/adenomas. | When available the histological report of polyps removed (up to 3 weeks).
  The percentage of adenomas, polyps (in general), flat adenoma and serrated polyps/adenoma detected will be recorded and compared between the groups.
Size of lesions detected | Immediately after the procedure.
  The size of lesion detected will be measured in millimiters and compared between the groups.
Rate of neoplasia by colonic site | Immediately after the procedure.
  The percentage of patients with neoplasia of proximal (right colonic segments) or distal (left colonic segments and rectum) site will be assessed and compared between the groups.
Post-colonoscopy surveilance | When available the histological report of polyps removed (up to 3 weeks).
  the time interval, expressed in years, to the next suggested follow-up colonoscopy will be assessed and compared between the groups.
Time of cecal intubation. | Immediately after the procedure.
  The time to reach the cecum will be measured in minutes, recorded and compared between the groups.
Withdrawal and total procedure time. | Immediately after the procedure.
  The time of withdrawal (from cecum to anus) and of the overall colonoscopy (from anus to anus) will be measured in minutes, recorded and compared between the groups.
Learning curve. | 3, 6, 9 and 12 months.
  The above-mentioned outcomes will be calculated for each endoscopist at 3, 6, 9 and 12 months.
Specific contribution of AI | Immediately after the procedure.
  Proportion of patients diagnosed with polyps which were detected only by Artificial intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Cristiano Spada, Principal Investigator — Fondazione Poliambulanza
Locations (1):
- Fondazione Poliambulanza, Brescia, Bs, Italy

IPD SHARING:
Plan to Share IPD: No